CLINICAL TRIAL: NCT02784119
Title: APCext : Effect of Temporary Porto-caval Shunt During Liver Transplantation on Function of Liver Graft From Extended Criteria Donor
Acronym: APCext
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2016-A00612-49; 35RC15_8975 (Other: CHU Rennes)
Record Dates: First submitted 2016-05-19; First posted 2016-05-26 (Estimated); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Liver Transplantation
Keywords: temporary porto-caval shunt; liver graft; extended criteria donor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- temporary porto-caval shunt (Experimental): patients in whom temporary porto-caval shunt is performed during orthotopic liver transplantation
  Interventions: Procedure: temporary porto-caval shunt
- no temporary porto-caval shunt (No Intervention): patients in whom temporary porto-caval shunt is not performed during orthotopic liver transplantation

INTERVENTIONS:
Procedure: temporary porto-caval shunt — temporary porto-caval shunt
  Arms: temporary porto-caval shunt

SUMMARY:
The success of orthotopic liver transplantation (OLT) in treatment of liver malignancy and endstage liver disease has led to an increase in the gap between patients on waiting-lists and available liver grafts. In order to compensate for this scarcity, use of liver grafts harvested from extended criteria donors (ECD) has become more and more frequent.

However, these ECD grafts are known to be associated with a higher rate of primary non function (PNF) or early allograft dysfunction (EAD) because of a greater vulnerability to ischemia-reperfusion injury (IRI).

During OLT, the clamping of the portal vein induces blood congestion in the splanchnic territory leading to increased gut permeability, bacterial translocation and release of endotoxin and pro-inflammatory cytokines at revascularisation, which exacerbate IRI.

Realisation of a temporary porto-caval shunt (TPCS) (i.e. end to side anastomosis between the portal vein and infrahepatic vena cava) during the anhepatic phase, avoids splanchnic congestion and could therefore decrease IRI and improve liver graft function. However, TPCS remains poorly used as no randomised trial succeeds to show its benefit on liver function due to lack of power.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Candidate of liver transplantation
* With cirrhosis from any etiology
* Model For End-Stage Liver Disease (MELD) score < 25
* Transplanted with a liver graft harvested from an extended criteria donor defined as presence of at least one of the following criteria:

  * Donor age > 65 years old
  * Intensive care unit stay > 7 days
  * BMI > 30
  * Natremia > 155 mmol/L
  * Aspartate aminotransferase (ASAT) > 150 IU/mL
  * Alanine aminotransferase (ALAT) > 170 IU/mL
  * Occurrence of a cardiac arrest before graft harvesting
  * Proven biopsy macrosteathosis > 30%
* Non-opposition from the patient

Non Inclusion Criteria:

* Fulminant hepatitis
* Retransplantation
* Combined organ transplantation (kidney, pancreas, heart, lung)
* Non heart beating donor
* Complete portal vein thrombosis on preoperative imaging finding

Exclusion Criteria:

* Complete portal vein thrombosis found during procedure
* Split liver graft
* Realisation of a bilio-enteric anastomosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2017-03-28 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of early allograft dysfunction | on postoperative day 7
  defined by the presence of at least one of the following criteria:
  * Bilirubin level > 10 mg/dL (i.e. 171 µmol/L)
  * International Normalized Ratio > 1.6
Incidence of early allograft dysfunction | within the 7 first postoperative day
  defined by the presence of at least one of the following criteria:
  • ASAT or ALAT level > 2000 IU/mL
Incidence of primary non function | within the 7 first postoperative day
  defined by the presence of at least one of the following criteria:
  * Graft's death or retransplantation
  * Patient's death

SECONDARY OUTCOMES:
Realisation of intra-operative transfusion | during the operation
  defined by the transfusion needs of fresh frozen plasma, red blood cell and platelet pool
Incidence of reperfusion syndrome | during the 5 minutes following revascularisation
  defined as decrease of 30% of the median arterial pressure
Duration of surgery | at day 0
Liver graft function | within 3 months
  evaluated by the Model for Early Allograft Function (MEAF) score
Occurrence of a severe postoperative complication | within 3 months
  defined as a Clavien-Dindo classification > 2
Evaluation of urinary function | within the first 7 days
  defined by:
  * Measuring postoperative creatinine level (mg/L)
  * Need of renal dialysis
Graft's survival | at 3 months
  defined by graft's death or retransplantation
Patient's survival | at 3 months
  defined by patient's death

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CHU Bordeaux, Bordeaux
  - Hospices Civils Lyon, Lyon
  - CHU Nice, Nice
  - CHU Rennes, Rennes
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours